CLINICAL TRIAL: NCT01950351
Title: Phase II Trial of Hypofractionated Proton Beam Therapy in Men With Localized Prostate Adenocarcinoma
Brief Title: Hypofractionated Proton Beam Therapy for Localized Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-1003; NCI-2013-02347 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-1003 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Stage I Prostate Adenocarcinoma AJCC v7; Stage II Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — Proton Therapy; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (proton beam radiation therapy) (Experimental): Patients undergo proton beam radiation therapy in 15 fractions over 5-6 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Proton Beam Radiation Therapy — Undergo proton beam radiation therapy
  Other Names: PBRT; Proton Radiation Therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies the side effects and how well hypofractionated proton beam radiation therapy works in treating patients with prostate cancer that has not spread to nearby lymph nodes or to other parts of the body. Specialized radiation therapy, such as proton beam radiation therapy, that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the incidence of grade 2 gastrointestinal toxicity following the proposed treatment regimens at 2 years post-treatment.

SECONDARY OBJECTIVES:

I. Estimate the change in health related quality of life (HRQOL) following the proposed treatment regimen compared to pre-treatment assessment as defined by Expanded Prostate Cancer Index Composite (EPIC), Utilization of Sexual Medications/Devices, and Medical history/conditions questionnaire.

II. Estimate the rates of acute toxicity of the treatment regimens. III. Estimate the rates of late toxicity at 3, 4, and 5 years post-treatment. IV. Assess the efficacy of hypo-fractionated proton beam therapy, defined by the incidence of a rising prostate-specific antigen (PSA) at 5 years.

V. Determine the rate of local failure by biopsy of the prostate when objective tests, prostate-specific antigen (PSA), magnetic resonance imaging (MRI), digital rectal exam (DRE), suggest relapse.

OUTLINE:

Patients undergo proton beam radiation therapy in 15 fractions over 5-6 weeks.

After completion of study treatment, patients are followed up every 6-12 months for 24 months and then annually until month 60.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate within one year of study entry; evaluation can happen outside of MD Anderson as long as histological confirmation takes place at MD Anderson
* History/physical examination with digital rectal examination of the prostate within 90 days prior to registration
* Histological evaluation of prostate biopsy with assignment of a Gleason score to the biopsy material demonstrating Gleason score 2-7 within 365 days of registration
* Clinical stage T1-2b (American Joint Committee on Cancer [AJCC] 7th edition) and PSA < 20 ng/mL within 90 days prior to registration; PSA should not be obtained within 10 days after prostate biopsy
* Zubrod performance status 0-1 within 90 days prior to registration
* Patient must be able to provide study-specific informed consent prior to study entry
* Willingness and ability to complete the EPIC questionnaire

Exclusion Criteria:

* Prior or concurrent invasive malignancy (except non-melanomatous skin cancer or lymphomatous/hematogenous malignancy) unless continually disease free for a minimum of 5 years
* Evidence of distant metastases
* Regional lymph node involvement
* Previous prostatectomy, cryosurgery, or high intensity focused ultrasound (HIFU) for prostate cancer
* Previous pelvic radiation or prostate brachytherapy
* Active and severe medical co-morbidity defined as follows: unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months, transmural myocardial infarction within the last 6 months, acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration, chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration, hepatic insufficiency resulting in clinical jaundice, active inflammatory bowel disease (Crohn's disease or ulcerative colitis), diagnosed connective tissue disorder, or congenital coagulation defects (patients on medical therapy with Coumadin or other blood thinning agents are eligible for participation)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of late grade 2 or greater gastrointestinal (GI) toxicity | Up to 2 years post-treatment
  The cumulative incidence of late grade 2 or greater GI toxicity will be estimated with a 95% confidence interval.

SECONDARY OUTCOMES:
Rates of acute toxicity | Within 90 days of treatment initiation
  Rates of acute toxicity will be assessed.
Rate of late toxicity | Up to 5 years post-treatment
  Rate of late toxicity will be determined.
Change in health related quality of life (HRQOL) as assessed by the Expanded Prostate Cancer Index Composite (EPIC) Utilization of Sexual Medications/Devices, and Medical history/conditions questionnaire | Baseline to up to 5 years
  Change in HRQOL will be evaluated.
Incidence of rising prostate-specific antigen (PSA) | At 5 years
  Incidence of rising PSA will be assessed.
Rate of local failure by biopsy | Up to 5 years
  Rate of local failure by biopsy will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Frank, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org